CLINICAL TRIAL: NCT00668122
Title: Efficacy and Safety of Ciprofloxacin Extended-Release 1000 mg Once-Daily Versus Ciprofloxacin Immediate-Release 500 mg Twice-Daily Given 7-14 Days in Patients With Complicated Urinary Tract Infections: Prospective, Randomized, Double-Blind Trial.
Brief Title: Efficacy and Safety of CIPRO XR Versus CIPRO IR in Patients With Complicated Urinary Tract Infections
Acronym: EMERON
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Therapeutic Area Head, Bayer HealthCare AG
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11454
Record Dates: First submitted 2008-04-24; First posted 2008-04-28 (Estimated); Last update posted 2009-06-30 (Estimated); Status verified 2009-06

CONDITIONS: Urinary Tract Infection
MeSH Terms: conditions — Urinary Tract Infections | interventions — Ciprofloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Cipro XR (Ciprofloxacin, BAYQ3939)
- Arm 2 (Experimental)
  Interventions: Drug: Cipro IR (Ciprofloxacin, BAYQ3939)

INTERVENTIONS:
Drug: Cipro XR (Ciprofloxacin, BAYQ3939) — Ciprofloxacin XR 1000 mg orally once a day
  Arms: Arm 1
Drug: Cipro IR (Ciprofloxacin, BAYQ3939) — Ciprofloxacin IR 500 mg orally twice a day
  Arms: Arm 2

SUMMARY:
To assess and compare the efficacy and safety of ciprofloxacin extended-release (CIPRO XR) tablet 1000 mg PO once-daily (OD) versus ciprofloxacin immediate-release (CIPRO IR) tablet 500 mg PO twice-daily (BID) for 7-14 days in patients with complicated and/or nosocomial urinary tract infections (cUTI).

ELIGIBILITY:
Inclusion Criteria:

The primary diagnosis in this clinical trial was cUTI in men or non-pregnant women over 18 years of age. Other main inclusion criteria:

* One or more clinical symptoms and signs of a lower UTI: fever (> 38°C, orally), chills, frequency of micturition, dysuria, urge sensation.
* One or more of the following underlying conditions suggestive of cUTI:
* Indwelling urinary catheter.
* 100 mL of residual urine after voiding.
* Neurogenic bladder.
* Obstructive uropathy due to lithiasis, tumor or fibrosis.
* Acute urinary retention in men.

Exclusion Criteria:

Diagnosis of pyelonephritis supported by clinical signs/symptoms of fever (>38°C orally), chills and flank pain (all 3 signs/symptoms must be present).

* Have a history of allergy to quinolones
* Are unable to take oral medication
* Have an intractable infection requiring > 14 days of therapy
* Have a requirement for concomitant administration of sucralfate or divalent and trivalent cations such as iron or antacids containing magnesium, aluminum or calcium
* Have prostatitis or epididymitis
* Have had a renal transplant
* Have ileal loop or vesica- urethral reflux
* Have significant liver or kidney impairment
* Have a history of tendinopathy associated with fluoroquinolones
* Are pregnant, nursing
* Have a history of convulsions or CNS disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2004-03; Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Bacteriological response 5 to 9 days after the last dose of study medication (TOC visit). | 5-9 days

SECONDARY OUTCOMES:
Bacteriological outcome during treatment | 7-14 days
Bacteriological outcome at follow-up | 28-42 days
Clinical outcome during treatment | 7-14 days
Clinical outcome at the test-of-cure visit | 5-9 days
Clinical outcome at follow-up | 28-42 days
Adverse event collection | 28-42 days

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (35):
- Italy (35):
  - Monza, Milano
  - Camposampiero, Padova
  - Orbassano, Torino
  - Busto Arsizio, Varese
  - Bassano del Grappa, Vicenza
  - Alessandria
  - Bari
  - Benevento
  - Bergamo
  - Bologna
  - Caserta
  - Catania
  - Chieti
  - Florence
  - Frosinone
  - Genova
  - L’Aquila
  - Mantova
  - Massa Carrara
  - Messina
  - Milan
  - Napoli
  - Palermo
  - Perugia
  - Potenza
  - Reggio Calabria
  - Reggio Emilia
  - Rimini
  - Roma
  - Sassari
  - Syracuse
  - Torino
  - Trieste
  - Varese
  - Verona